CLINICAL TRIAL: NCT07238543
Title: Comparative Study of Novel Prognostic Scores for Prediction of Morbidity and Mortality in Patients With Liver Cirrhosis
Brief Title: Comparative Study of Novel Prognostic Scores in Patients With Liver Cirrhosis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Hany Youssef Mina, Dr, Assiut University
Other Study IDs: New scores in liver cirrhosis
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Usage of new scores — usage of new scores for prediction of morbidity and mortality in patients with liver cirrhosis

SUMMARY:
1. To determine the prognostic performance of novel scores in predicting complications and in-hospital mortality in patients with liver cirrhosis.
2. To compare the accuracy of these scores in identifying high risk patients relative to the standard scores.

DETAILED DESCRIPTION:
* Liver cirrhosis represents the end stage of chronic liver diseases and remains a major global health burden, accounting for over 1 million deaths annually.
* It is characterized by progressive fibrosis, nodular regeneration, and architectural distortion of the liver parenchyma, ultimately leading to liver dysfunction and portal hypertension
* Once acute decompensation occurs the prognosis significantly worsens, with a sharp increase in short-term mortality
* Accurate outcome prediction in cirrhotic patients is essential for guiding early interventions, allocating healthcare resources, and prioritizing liver transplant listing.
* Traditional prognostic scores, such as the Child-Turcotte Pugh (CTP) and Model for End-Stage Liver Disease (MELD), have important limitations.
* CTP includes subjective variables, while MELD may not fully reflect clinical deterioration in early decompensation
* MELD is widely used to predict the short-term mortality in patients with cirrhosis, but potential limitations of this score have been reported.
* An integrated MELD model (iMELD) including serum sodium and age improves the prediction of early mortality in patients with cirrhosis The Chronic Liver Failure Consortium Acute Decompensation (CLIF-C AD) score, introduced by European Association for the Study of the Liver (EASL), was specifically designed for hospitalized patients with acute decompensation (without Faculty of Medicine Institutional Review Board (IRB) Assiut Medical School Research Proposal Form 3 ACLF). It incorporates age, white blood cell count, and organ function to better stratify risk
* Recently, newer prognostic models such as the ADRECIA score have been developed, incorporating variables such as inflammatory markers and kidney function. These models aim to further refine risk stratification in cirrhosis, especially in early decompensation, before organ failure sets in
* Although these novel scores show promise in identifying patients at high risk for deterioration or death, direct comparisons in real-world clinical settings are lacking.
* Understanding their relative performance could help optimize the management of hospitalized patients with AD cirrhosis, thereby facilitating early clinical decision-making, optimizing patient outcomes, and potentially improving resource allocation in hepatology care settings.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years

  * Diagnosis of liver cirrhosis (clinical, radiological using ultrasound or fibroscan)
  * Hospital admission for acute decompensation (ascites, hepatic encephalopathy, variceal bleeding, SBP)

Exclusion C• Previous liver transplantation

* Pregnancy
* Refusal to participate in the study riteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study based on patients with Liver Cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Comparative study of novel prognostic scores for prediction of morbidity and mortality in patients with liver cirrhosis | baseline
  Usage of new prognostic scores for prediction of morbidity and mortality in patients with LC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jalan R, Saliba F, Pavesi M, Amoros A, Moreau R, Gines P, Levesque E, Durand F, Angeli P, Caraceni P, Hopf C, Alessandria C, Rodriguez E, Solis-Munoz P, Laleman W, Trebicka J, Zeuzem S, Gustot T, Mookerjee R, Elkrief L, Soriano G, Cordoba J, Morando F, Gerbes A, Agarwal B, Samuel D, Bernardi M, Arroyo V; CANONIC study investigators of the EASL-CLIF Consortium. Development and validation of a prognostic score to predict mortality in patients with acute-on-chronic liver failure. J Hepatol. 2014 Nov;61(5):1038-47. doi: 10.1016/j.jhep.2014.06.012. Epub 2014 Jun 17. PMID 24950482
- [Result] Asrani SK, Devarbhavi H, Eaton J, Kamath PS. Burden of liver diseases in the world. J Hepatol. 2019 Jan;70(1):151-171. doi: 10.1016/j.jhep.2018.09.014. Epub 2018 Sep 26. PMID 30266282